CLINICAL TRIAL: NCT04018404
Title: Family Resilience Initiative Research Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LB_FRI RESEARCH
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Adverse Childhood Experiences

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Subjects will be approached for enrollment prior to or following clinic visit with physician. Only children present with a biological mother will be considered for enrollment. Charts of controls will be flagged so that they will not be able to be enrolled in the FRI clinical program if they present to a morning clinic where the program is offered.
- Subject (Experimental): Mothers and children will be approached by study personnel (separate from Outreach Coordinators who will obtain consent for use of information to evaluate the FRI Clinical Program) for enrollment in the FRI Research Program following completion of all FRI Clinical Program activities for that day. Both mother and child will be enrolled and contribute data and samples to the FRI Research Program.
  Interventions: Other: FRI CLINICAL PROGRAM

INTERVENTIONS:
Other: FRI CLINICAL PROGRAM — University Le Bonheur Pediatric Specialists and Le Bonheur Community Health and Well-Being, Maternal Child Department, have started the Family Resilience Initiative (FRI) in the ULPS General Pediatrics Clinic. This clinical program screens children 9 months to less than five years of age for ACES and SDH at the time of presentation for well child checks. There are two outreach coordinators who screen and enroll children attending clinic for a well-child check during morning clinics 3 to 4 days per week. Children with positive screens for ACES and/or SDH, and their adult caregivers, receive community resource referrals with warm handoffs to vetted organizations. In addition, if indicated, psychological services are offered for children based upon the presence of one or more of ACEs and current health and behavioral problems.
  Arms: Subject

SUMMARY:
University Le Bonheur Pediatric Specialists (ULPS) and Le Bonheur Community Health and Well-Being, Maternal Child Department, have started the Family Resilience Initiative (FRI) in the ULPS General Pediatrics Clinic. This clinical program screens children 9 to 48 months of age for Adverse Childhood Experiences (ACEs) and Social Determinants of Health (SDH) at the time of presentation for well child checks. Children with positive screens for ACES and/or SDH, and their adult caregivers, receive community resource referrals with warm handoffs to vetted organizations. In addition, if indicated, psychological services are offered for children based upon the presence of one or more of ACEs and current health, social, and behavioral problems. It is expected that enrollment in FRI will improve quality of life for families through reduction in stress by addressing unmet social needs and providing psychological counseling of children and families with any ACE exposure. The investigators expect that FRI will have a positive impact on the physical health, healthcare utilization, mental health, development, and school readiness of children in the program compared to controls. The investigators will compare changes in weight for height and blood pressure percentiles at enrollment and end of study and the number of unscheduled healthcare visit for illness for children in the FRI clinical program compared to controls, receiving standard of care. Healthcare visits include visits to the clinic and visits to the Le Bonheur Emergency Department. The investigators will also compare pre- and post-treatment scores on the validated Child Behavior Checklist and Parenting Stress Index as a measure of stress reduction. Furthermore, the investigators will measure age appropriate attainment of developmental milestones scores on early, school-based testing (MAP) testing scores obtained through Seeding Success. The investigators will also determine rates of physician-diagnosed early behavioral disorders such as ADHD. The investigators expect that reduced stress and its downstream conditions will lead to decreased healthcare visits, improved attainment of developmental and educational milestones, and lower rates of behavioral disorders.

DETAILED DESCRIPTION:
Adverse childhood experiences (ACEs), social determinants of health (SDH) and their downstream health effects are the public health crisis of our time. Many chronic diseases are known to originate with, or are exacerbated by, exposure to toxic stress in childhood including learning and cognitive disabilities, asthma, obesity, diabetes, cancer, and behavioral health disorders such as ADHD, depression and substance abuse. While poverty is not considered an ACE, ACE exposure and unmet social needs are more common in those living in lower income communities. Memphis, the poorest statistical metropolitan area in the country with a population over one million people has an overall poverty rate of 26.9% and a child poverty rate of 44.7%. A telephone survey of over 1500 Shelby County residents conducted in the summer of 2014 found that 52% of adults reported at least one ACE and 12% reported four or more. Race is also an important factor in health disparities. Although the effects of race are predominantly due to associated income inequities, systemic racism can also have effects on health. For example, disparities in birth outcomes between black and white mothers exists across all socioeconomic strata but is most prominent among highly educated African American women.

The association between poverty and ill health is likely mediated through several pathways. In impoverished households there may be limited cognitive stimulation and neglect. Poor quality and location of housing may expose children to environmental toxins such as lead or air pollution and allergens. Poor diet may result in micronutrient deprivation. In addition to these known negative exposures, environmental stress through exposure to familial discord and disruption, intrafamily violence, overcrowding of the home, and neighborhood violence appears also to play a role in the poor mental and physical health of individuals with these exposures.

The link between toxic stress from ACES and other social determinants of health and adverse physical and mental health outcomes is derived from mostly cross-sectional studies where individuals with and without certain health conditions are compared for exposure to ACEs and SDH. These studies have been critical in revealing the spectrum of childhood and adult conditions that may be triggered or exacerbated by toxic stress. Both acute severe stress stemming from exposures like child maltreatment and chronic lower grade stresses stemming from exposure to poverty and its associated risks are associated with physical and mental illness. Much of the research into the mechanisms underpinning these associations has examined the epigenetic effect of these episodic or longer-term stressors. Epigenetics refers to post-translational modifications of DNA such as methylation, the covalent binding of methyl groups at CpG sites, oligodeoxynucleotides where cytosine is adjacent to guanine. Changes in methylation patterns can result from de novo methylation of DNA or removal of pre-existing methylation sites. Most epigenetic changes influence gene transcription through methylation of promotor and repressor regions. A gene promotor containing methylated CpG sequences is less able to bind transcription factors resulting in reduced gene transcription. Many studies have found differential methylation of areas within genes as well as intergenic areas of DNA. The effect these areas of methylation have on gene expression are unknown. Histones, proteins around which DNA is coiled, can be modified as well through methylation and acetylation. These modifications are thought to relax DNA coiling and open up gene regulatory sites for interaction with transcription factors.

There have been studies examining differences in methylation across the genome, comparing the number of sites with increased and reduced methylation and drawing inferences as to the effect of these differences on phenotype. Many such studies have demonstrated clear differences in methylation patterns between subjects with greater and lesser exposure to episodic and lifetime stress. Differential methylation of specific genes and their promotor regions have also been studied, specifically, genes that could be reasonably hypothesized to play a role in the response to stress and the mitigating effects of different levels of caregiving. These include the genes for the glucocorticoid receptor, serotonin and oxytocin. The effects of chronically or acutely elevated cortisol levels on the methylation of the glucocorticoid receptor gene and its promotor are, perhaps, the most extensively studied in relation to ACEs and SDH. Animal studies have demonstrated an effect of high levels of caregiving on levels of glucocorticoid receptor expression in key areas of the brain through epigenetic changes which can improve self-regulation and mitigate the effects of toxic stress. These epigenetic modifications have been demonstrated to be transmitted across generations and may account for cross generational protection or vulnerability to the effects of toxic stress.

Most human data on the effects of epigenetics are derived from retrospective and cross-sectional studies in which individuals with certain health conditions report on past or current exposure to ACEs and/or SDH. Many of these studies examine the cumulative risk of exposure over the lifetime of the study subject up to the point of the research. There does appear to be a dose response relationship between earlier stressors and adolescent and adult mental and physical health. Interventions applied early may, therefore, have the potential to mitigate the effects of toxic stress on health even if exposures have already occurred and prevent these important, long-term impacts on health and well-being. Mitigating factors include high family functioning with lower levels of parental stress and greater parent-child communication, as well as access to a medical home.

Primary care is the cornerstone for screening, health promotion and disease prevention and pediatricians are best situated to screen for and address ACEs and SDH. Studies have demonstrated that many physicians do not perform any formal screening for ACEs but that individuals and families, when approached in a family-centered manner, want their physicians to screen for stressors and unmet social needs, even though it involves answering sensitive questions.

ELIGIBILITY:
Inclusion Criteria: Experimental group

- 1. Children born at 32 weeks or greater between the ages of 18 to 36 months and their biological mothers.

2. Present to a morning ULPS General Pediatric clinic for a well-child check and newly enrolled that day into the FRI Clinical program (requires at least one ACE or SDH disclosed on screening of child and agrees to clinical program) 3. Mother English speaking

Exclusion Criteria:

* 1. Previously enrolled in FRI Clinical Program 2. Previously enrolled as a control in an afternoon clinic 3. Previously identified serious chronic health problems (e.g. complex congenital heart disease)

Inclusion Criteria: Control group

1. Children born at 32 weeks or greater between the ages of 18 to 36 months and their biological mothers.
2. Presenting to an afternoon ULPS General Pediatric clinic for a well- child check
3. Has at least one ACE or SDH on pre-enrollment screening
4. Mother English speaking

Exclusion Criteria:

4. Previously enrolled in FRI Clinical Program 5. Previously identified serious chronic health problems (e.g. complex congenital heart disease)

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in CBCL score (behavioral measure) | after 3 years
  We will use the CBCL scores (total, internalizing and subscales, externalizing and subscales) to define behavior problems. Since we expect a high rate of loss to follow up during the study, we plan to recruit 195 subjects in each arm to account for up to 50% loss to follow up. Our target population for the primary outcome will therefore be 390.
Changes in BMI from baseline | after 3 years
  We will use changes in BMI to classify child as underweight, normal weight, overweight, obese.
Change in blood pressure percentile from baseline (health measure) | after 3 years
  We will use changes in blood pressure percentile to determine presence of hypertension.
Rate of diagnosis of ADHD (behavioral measure) | after 3 years
  We will use the diagnosis of ADHD to define specific behavioral problems
Percentiles on ASQ domains (developmental measure) | after 3 years
  We will use percentiles on ASQ domains to determine achievement of appropriate developmental milestones.
Measures of Academic Progress testing score (school age) | after 3 years
  Using the RIT (Rasch Units) to chart the students academic growth from year to year. Will be available once child has entered school and will be used to determine school readiness.
Change in Parenting Stress Index score (mother) | after 3 years
  We will use Parenting Stress Index to determine the level of parental stress. The PSI 120 item inventory that focuses on three major domains of stress (child characteristics, parent characteristics, and situational/demographic life stress.
Change in flourishing score (mother) | after 3 years
  This scale is used around the world to assess various domains of flourishing, or human well being. We will use changes in flourishing score to determine maternal well being

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing plan is to share data with other researchers as well as The IRB at the University of Tennessee Health Science Center, Le Bonheur Children's Hospital, UT Le Bonheur Pediatric Specialists, Inc., and Urban Child Institute which sponsors and provides funds for this research.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Until the study is complete
Access Criteria: The data will only be given to others to do the research, to study the results, and to see if the research was done correctly.

REFERENCES:
- [Background] Beck AF, Klein MD. Moving From Social Risk Assessment and Identification to Intervention and Treatment. Acad Pediatr. 2016 Mar;16(2):97-8. doi: 10.1016/j.acap.2016.01.001. Epub 2016 Jan 11. No abstract available. PMID 26791277
- [Background] Bick J, Naumova O, Hunter S, Barbot B, Lee M, Luthar SS, Raefski A, Grigorenko EL. Childhood adversity and DNA methylation of genes involved in the hypothalamus-pituitary-adrenal axis and immune system: whole-genome and candidate-gene associations. Dev Psychopathol. 2012 Nov;24(4):1417-25. doi: 10.1017/S0954579412000806. PMID 23062307
- [Background] Bright MA, Knapp C, Hinojosa MS, Alford S, Bonner B. The Comorbidity of Physical, Mental, and Developmental Conditions Associated with Childhood Adversity: A Population Based Study. Matern Child Health J. 2016 Apr;20(4):843-53. doi: 10.1007/s10995-015-1915-7. PMID 26694043
- [Background] Bright MA, Thompson L, Esernio-Jenssen D, Alford S, Shenkman E. Primary Care Pediatricians' Perceived Prevalence and Surveillance of Adverse Childhood Experiences in Low-Income Children. J Health Care Poor Underserved. 2015 Aug;26(3):686-700. doi: 10.1353/hpu.2015.0080. PMID 26320905
- [Background] Chung EK, Siegel BS, Garg A, Conroy K, Gross RS, Long DA, Lewis G, Osman CJ, Jo Messito M, Wade R Jr, Shonna Yin H, Cox J, Fierman AH. Screening for Social Determinants of Health Among Children and Families Living in Poverty: A Guide for Clinicians. Curr Probl Pediatr Adolesc Health Care. 2016 May;46(5):135-53. doi: 10.1016/j.cppeds.2016.02.004. Epub 2016 Apr 18. PMID 27101890
- [Background] Denhardt DT. Effect of stress on human biology: Epigenetics, adaptation, inheritance, and social significance. J Cell Physiol. 2018 Mar;233(3):1975-1984. doi: 10.1002/jcp.25837. Epub 2017 Apr 27. PMID 28158904
- [Background] Gottlieb L, Hessler D, Long D, Amaya A, Adler N. A randomized trial on screening for social determinants of health: the iScreen study. Pediatrics. 2014 Dec;134(6):e1611-8. doi: 10.1542/peds.2014-1439. Epub 2014 Nov 3. PMID 25367545
- [Background] Gottlieb LM, Hessler D, Long D, Laves E, Burns AR, Amaya A, Sweeney P, Schudel C, Adler NE. Effects of Social Needs Screening and In-Person Service Navigation on Child Health: A Randomized Clinical Trial. JAMA Pediatr. 2016 Nov 7;170(11):e162521. doi: 10.1001/jamapediatrics.2016.2521. Epub 2016 Nov 7. PMID 27599265
- [Background] Gottlieb LM, Wing H, Adler NE. A Systematic Review of Interventions on Patients' Social and Economic Needs. Am J Prev Med. 2017 Nov;53(5):719-729. doi: 10.1016/j.amepre.2017.05.011. Epub 2017 Jul 5. PMID 28688725
- [Background] Jimenez ME, Wade R Jr, Lin Y, Morrow LM, Reichman NE. Adverse Experiences in Early Childhood and Kindergarten Outcomes. Pediatrics. 2016 Feb;137(2):e20151839. doi: 10.1542/peds.2015-1839. Epub 2016 Jan 14. PMID 26768347
- [Result] Argentieri MA, Nagarajan S, Seddighzadeh B, Baccarelli AA, Shields AE. Epigenetic Pathways in Human Disease: The Impact of DNA Methylation on Stress-Related Pathogenesis and Current Challenges in Biomarker Development. EBioMedicine. 2017 Apr;18:327-350. doi: 10.1016/j.ebiom.2017.03.044. Epub 2017 Apr 4. PMID 28434943